CLINICAL TRIAL: NCT05226351
Title: Activation of the Endocannabinoid System and Cognition (Effekte Einer Akuten Aktivierung Des Cannabinoid-Systems Auf Kognitive Funktionen)
Brief Title: Activation of the Endocannabinoid System and Cognition
Acronym: DronaMemo-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Stefan Roepke, Prof. Dr. Stefan Röpke, Charite University, Berlin, Germany
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: WI 3396/14-1 // RO 3935/7-1
Record Dates: First submitted 2021-04-29; First posted 2022-02-07 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-08

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dronabinol PTSD (Active Comparator): Donabinol before cognitve testing - PTSD patients
  Interventions: Drug: Dronabinol 2.5 mg
- Dronabinol healthy controls (Active Comparator): Donabinol before cognitve testing - healthy controls
  Interventions: Drug: Dronabinol 2.5 mg
- Placebo PTSD (Placebo Comparator): Placebo before cognitve testing - PTSD patients
  Interventions: Drug: Placebo
- Placebo healthy controls (Placebo Comparator): Placebo before cognitve testing - healthy controls
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol 2.5 mg — single administration of 2.5mg Dronabinol oral (oily solution)
  Arms: Dronabinol PTSD; Dronabinol healthy controls
Drug: Placebo — single administration of placebo oral (oily solution)
  Arms: Placebo PTSD; Placebo healthy controls

SUMMARY:
Recent data suggest that the cannabinoid-system is involved in stress regulation and posttraumatic stress disorder (PTSD). Low endocannabinoid signaling has been found in PTSD patients and might even present a precondition to develop PTSD after trauma. The aim of the current project is to investigate the impact of an activation of the cannabinoid system with an exogenous cannabinoid (dronabinol, i.e., delta-9-tetrahydrocannabinol) on fear conditioning.

DETAILED DESCRIPTION:
Recent data suggest that the cannabinoid-system is involved in stress regulation and posttraumatic stress disorder (PTSD). Low endocannabinoid signaling has been found in PTSD patients and might even present a precondition to develop PTSD after trauma. In consequence, increased endocannabinoid signaling during acquisition and consolidation of traumatic events might be a promising approach to prevent the development of PTSD. The aim of the current project is to investigate the impact of an activation of the cannabinoid system with an exogenous cannabinoid (dronabinol, i.e., delta-9-tetrahydrocannabinol) on tfear conditioning in patients with PTSD and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* PTSD criteria fullfilled (patients only)

Exclusion Criteria:

* All cases of physical illnesses and intake of medication (except oral contraceptives) (healthy controls only) will be excluded.
* Pregnant and lactating individuals will also be excluded. Participants with a positive urinary cannabinoid test (Cannabis 20 Pipettier-Drogenschnelltest (Urin), Diagnostik Nord GmbH) will also be excluded.
* psychiatric disorder according to DSM-5 (healthy controls only)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
extinction learning | 30 minutes
  extinction learning in fear conditioning paradigm: skin conductance reaction

SECONDARY OUTCOMES:
empathy | 15 minutes
  cognitive and emotional empathy: number of correct answers & rating of own emotional state
Probabilistic Reversal Learning Task | 15 minutes
  learning and cognitive flexibility: reaction times
selective attention | 10 minutes
  emotional dot-probe task: attentional bias index

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Charité Universitätsmedizin Berlin, Berlin
  - Charite University, Berlin

IPD SHARING:
Plan to Share IPD: Undecided